CLINICAL TRIAL: NCT03836560
Title: Comparing the Effectiveness of Nicotine Patch With Gum Versus Nicotine Patch Alone in Smoking Cessation in Hong Kong Primary Care Clinics
Brief Title: Comparing the Effectiveness of Combined NRT With Single NRT in Primary Care Clinics in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Maria Leung, Consultant in Family Medicine, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HA_SCCP_NRT
Record Dates: First submitted 2019-01-30; First posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Smoking Cessation
Keywords: nicotine replacement therapy; smoking cessation; quit rates
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Intervention Model Description: One year, 2 arm, parallel, randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor did not know which arm was interventional/control during the data analysis process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual group (Active Comparator): Usual group with nicotine patch only:
  Usual care involved counseling and 8 weeks of single NRT of nicotine patch. For those smoking 20 or more cigarettes per day before quitting, the NRT patch regimen was 4 weeks of 21mg patches, then 2 weeks of 14mg patches, followed by 2 weeks of 7mg patches. For those smoking 10 to 19 cigarettes per day before quitting, the NRT patch regimen was 4 weeks of 14mg patches, followed by 4 weeks of 7mg patches.
  Interventions: Drug: Nicotine patch
- Intervention group (Active Comparator): Nicotine patch and nicotine gum:
  Intervention consisted of counseling and 8 weeks of combined NRT of nicotine patch and gum. For those smoking 20 or more cigarettes per day before quitting, the NRT patch regimen was 4 weeks of 21mg patches, then 2 weeks of 14mg patches, followed by 2 weeks of 7mg patches. For those smoking 10 to 19 cigarettes per day before quitting, the NRT patch regimen was 4 weeks of 14mg patches, followed by 4 weeks of 7mg patches. 2mg nicotine gum was used once every 1 to 2 hours when required.
  Interventions: Drug: Nicotine patch; Drug: Nicotine gum

INTERVENTIONS:
Drug: Nicotine patch — nicotine patch given for 8 weeks
Drug: Nicotine gum — nicotine gum given as requested
  Arms: Intervention group

SUMMARY:
The prevalence of cigarette smoking has dropped to 10% in Hong Kong (HK) in 2017, however, smoking still kills 5700 persons per year. Studies suggest that abstinence rates are higher with combined NRT than single NRT, although local data on safety and benefits of combined NRT are lacking.

This is a one-year, two-arm, parallel randomized trial in 20 HK public clinics. The aim is to compare the effectiveness of combined NRT with single NRT among HK Chinese. 560 chronic smokers, who smoked ≥10 cigarettes/day for ≥ 1 year, were randomized to either intervention or usual care.

Intervention group received counseling and nicotine patch & gum. Usual care group received counselling and nicotine patch only. Primary outcome was smoking abstinence rate at 52 weeks. Secondary outcomes included smoking abstinence rate at 4, 12, & 26 weeks. Crude odds ratio (combined NRT vs. single NRT) and p-value were reported from logistic regression without adjustment; for trend analysis, adjusted odds ratio (AOR) and p-value were reported from Generalized Estimating Equation (GEE) (controlling for time). All AORs were adjusted for age, sex, baseline CO and clusters.

DETAILED DESCRIPTION:
Background Globally, smoking causes six million deaths a year1. By 2030, if current trends continue, the number of deaths will rise to eight million. According to Hong Kong Thematic Household Survey Reports, although the prevalence of current smokers among aged 15 and over has dropped from 15.3% in 2006 to 10.8% in 2017 in Hong Kong, smoking still kills 5700 persons per year and contributes to 14% of all deaths from non-communicable diseases. Thus, enhancement in smoking cessation would be crucial in improving health all smokers.

Among all pharmacological treatment for smoking cessation, evidences showed that oral treatment such as Varenicline is the most clinically effective smoking cessation medication9. However, there have been concerns about its adverse effect on neuropsychiatric and cardiovascular aspects. Besides, many smokers are reluctant to use it due to fear of its high rate of side effects and being medicalized for smoking cessation. The use of nicotine replacement therapy (NRT) has been largely studied, and, over the last decade, many studies had been carried out to compare the effect of monotherapy with combined nicotine replacement therapy. While the effect of monotherapy had been found to be small in heavy smokers due to significant withdrawal symptoms, combined NRT is believed to provide a stable baseline nicotine level by means of nicotine patch plus intermittent usage of short acting NRT e.g. gums, lozenges or inhalers for withdrawal symptoms. Several studies have shown that combined NRT is associated with lower withdrawal scores and higher 6-month quit rates (26.9 to 36.9%) when compared with monotherapies (19-23%)18-21. Combined NRT has also been shown to be safe as trials of combining various NRTs did not report that combination treatment produced increased adverse events.

In Hong Kong, Hospital Authority is one of the major service providers for smoking cessation. The target recipients of our smoking cessation service are primarily patients attending public general out-patient clinics (GOPCs) for management of chronic illnesses such as hypertension and diabetes mellitus, as well as patients with episodic complaints. Through effective interventions provided in the smoking cessation service, it is aimed that their medical conditions could be further improved. However, as majority of these smokers have moderate or above nicotine dependence, how effective is combined NRT compared to single NRT in this Chinese population is unknown.

Hypothesis:

Combined NRT gives a higher abstinence rate than single NRT.

Objective:

This study aims to compare the effectiveness of combined NRT with single NRT in Hong Kong primary care clinics.

Assessment Patients were seen at baseline for assessment, and then at 4 weeks, 12 weeks, 26 weeks and 52 weeks. Study medication was given at baseline and at week 4. In baseline assessment, smoking history including daily cigarette consumption and past quitting method, past medical health, drug history and allergy would be obtained. In follow up visits patients were assessed on nicotine withdrawal symptoms, carbon monoxide level, side effects from treatment and medication compliance. Counselling would be given in all follow up visits.

Pharmacological interventions Patients were randomized to either intervention or usual care for smoking cessation. Nicotine replacement therapy (NRT) was given for 8 weeks in both arms. Intervention consisted of counseling and combined NRT of nicotine patch and gum. Usual care involved counseling and single NRT of nicotine patch. NRT patch regimen used in usual care was the same as that in intervention group.

Data analysis Baseline characteristics were reported and compared by treatment groups, two-sample t test was conducted for continuous variables and Chi-square test for categorical variables. At each visit, crude odds ratio (OR) (combined NRT vs. single NRT) was reported, simple logistic regression was utilized without adjustment first, and then adjusted for potential confounders, age, sex, baseline CO level and cluster site of the subject recruitment. The overall treatment effect (combined NRT vs. single NRT) over the study period was estimated by Generalized Estimating Equation (GEE). In the GEE model, time (repeated measures at 4, 12, 26, and 52 weeks) was included as a continuous covariate, adjusted odds ratio (AOR) was reported and treatment-time interaction was tested. Potential confounders were also adjusted for in the GEE model. As GEE only uses non-missing records, missing at complete random was assumed to avoid bias. To support the random missing assumption, supplementary analysis was conducted for missingness pattern Furthermore, imputation was conducted under a conservative scenario of 'all missing records as "failure", i.e., not quit'. Statistical significance level was set at two-sided p<0.05 for all tests. Analysis was conducted by R version 3.2.235. Side effects from NRT were also recorded from both groups. Chi-squared test was used to compare the difference.

ELIGIBILITY:
Inclusion Criteria:

* current smokers who smoke 10 or more cigarettes a day for at least one year

Exclusion Criteria:

* unstable angina
* severe cardiac arrhythmia
* recent acute myocardial infarction or cerebrovascular accident in preceding 3 months
* below 18 years old
* being pregnant or on breast-feeding
* unable to use gum
* with a previous history of failure to NRT
* with a history of hypersensitivity to nicotine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2012-12-18 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
7-day point-prevalence abstinence rate at 52 weeks after quit date | at 52 weeks after the agreed quit date
  During initial assessment, patient will set a quit date with the counsellor. At 52 weeks after the quit rate, counsellor will call the patient and confirm his quit status. The status was confirmed by self reporting abstinence rate and exhaled carbon monoxide level

SECONDARY OUTCOMES:
side effects profiles | up to 1 year
  side effects from nicotine replacement therapy
7-day point-prevalence of abstinence rate at 26 weeks after quit date | at 26 weeks after the agreed quit date
  During initial assessment, patient will set a quit date with the counsellor. At 26 weeks after the quit rate, counsellor will call the patient and confirm his quit status. The status was confirmed by self reporting abstinence rate and exhaled carbon monoxide level

CONTACTS AND LOCATIONS:
Overall Officials: David Chao, FHKAM, Study Chair — Hospital Authority

IPD SHARING:
Plan to Share IPD: Undecided
We plan to provide a dropbox link

REFERENCES:
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- [Derived] Leung MKW, Bai D, Yip BHK, Fong MY, Lai PMH, Lai P, Lai ISY, Lam ZHW, Leung ATF, To DKY, Wong MT, Wong TK, Chao DVK. Combined nicotine patch with gum versus nicotine patch alone in smoking cessation in Hong Kong primary care clinics: a randomised controlled trial. BMC Public Health. 2019 Oct 16;19(1):1302. doi: 10.1186/s12889-019-7634-z. PMID 31619205

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study protocol and statistical analysis plan (2012-12-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT03836560/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Results of the study (2018-11-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT03836560/Prot_SAP_001.pdf